CLINICAL TRIAL: NCT04909970
Title: Impact of a Self-hyPnOsis Practice on Chronic StresS Among Caregivers of Elderly People With Loss of Autonomy at Home: a Randomized Controlled Pilot Study With a Waiting List
Brief Title: Impact of a Self-hyPnOsis Practice on Chronic StresS Among Caregivers of Elderly People With Loss of Autonomy at Home
Acronym: POSSAID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/CHU/02
Record Dates: First submitted 2021-05-03; First posted 2021-06-02 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Stress
Keywords: Family caregivers; Aged persons; homebound persons; Chronic stress; Self-hypnosis
MeSH Terms: interventions — Hypnosis; Waiting Lists

STUDY DESIGN:
Intervention Model Description: waiting list
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self hypnosis (Experimental): Self-hypnosis program associated to usual practice of stress management
  Interventions: Other: Self-hypnosis
- control group (waiting list) (Other): Usual practice of stress management. This group will practice self-hypnosis after the intervention group has practiced self-hypnosis (waiting list).
  Interventions: Other: Control (Waiting list)

INTERVENTIONS:
Other: Self-hypnosis — Self-hypnosis training during 8 weeks and one daily self-hypnosis session during 8 weeks
  Arms: Self hypnosis
Other: Control (Waiting list) — Usual practice during the first 16 weeks. At the end of study, the participant will practice Self-hypnosis training during 8 weeks and one daily self-hypnosis session during 8 weeks
  Arms: control group (waiting list)

SUMMARY:
In France, stress particularly affects family caregivers because of the intensive help they provide on a permanent basis to people losing their autonomy at home. This care work is often considered as a "burden" and has all the characteristics of a chronic daily stress factor. The prevalence of stress among caregivers is high and the level of stress varies according to the type of care provided to seniors at home.

This chronic stress has harmful effects on the health of family caregivers (depression, fatigue, insomnia, onset of chronic diseases, early mortality). It can be detrimental to their well-being and quality of life.

However, ageing well at home for older people is based on this essential pillar: the caregivers. They must remain in good physical and psychological health. Reducing their daily stress is becoming a public health challenge and a national priority.

Currently, the management of caregiver stress is based on several measures and devices. Non-conventional care practices such as Mindfulness-Based Stress Reduction, meditation, relaxation and yoga are offered to family caregivers. Initial results of studies on the effect of these complementary medicines show an improvement in psychological stress. However, research in this field is relatively recent. The conclusions must therefore be approached with caution. Moreover, no medium or long-term evaluation has been found in the scientific literature.

Self-hypnosis is becoming a common practice in healthcare. It has demonstrated its effectiveness in reducing pain and anxiety in both adults and children. In addition, other recent scientific evidence supports the effectiveness of hypnosis in stress management. In France, no study on caregiver stress and its management by self-hypnosis has been identified in the literature. The hypothesis is that the stress level of caregivers of elderly people at home could be reduced through daily self-hypnosis practice at home.

ELIGIBILITY:
Inclusion Criteria:

* Stress > or = 3 evaluated by the analogic visual scale of CHAMOUX
* Caregiver at home for a person uper than 60 years old with a loss of autonomy and followed in geriatrics or in polyvalent medicine
* Daily help in at least one of the 3 spheres of the elderly activity
* Person providing care services for more than 2 years with the elderly
* Person who can read and write
* Person affiliated to a social security scheme
* Person who gives his oral express consent
* Person who lives in Reunion Island

Exclusion Criteria:

* Person with serious chronic disorder (cancer for example)
* Person with a contraindication to hypnosis (cognitive and psychiatric disorders or alcohol dependence)
* Person under specific treatment preventing them from performing the intervention consistently
* Person who has already practiced hypnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of the feasibility of a practice of self-hypnosis on reducing the stress of carers caring for the elderly at home compared to a control group with waiting list. | week 16 after enrollment
  Membership of program participants : number of session of self-hypnosis realized compared to proposed session.
  It will be considered sufficient if 80% of the participants carry out 2 individual sessions and 1 collective hypnosis session during the training and practice 80% of the self-hypnosis sessions at home.
Assessment of the feasibility of a practice of self-hypnosis on reducing the stress of carers caring for the elderly at home compared to a control group with waiting list. | 6 months after the first enrollment
  number of patients recruited over 6 months Recruitment will be deemed acceptable if 60 participants are recruited over 6 months.

SECONDARY OUTCOMES:
Comparison of the variation in caregiver burden between inclusion and the end of self-hypnosis practice between the 2 groups of participant | week 16 after enrollment
  The burden will be evaluated by the Zarit scale min score = 0 and max score =88 score>60 = serious burden
Comparison of the variation in caregiver sleep quality between inclusion and the end of selfhypnosis practice between the 2 groups of participant | week 16 after enrollment
  The quality of sleep will be evaluated by the Pittsburgh Sleep Quality Index (PSQI) min score = 0 and max score = 32 score = 32 : extreme fatigue
Comparison of the variation in caregiver fatigue level between inclusion and the end of self-hypnosis practice between the 2 groups of participant | week 16 after enrollment
  The level of fatigue will be evaluated by the Pichot scale
Comparison of the variation in caregiver quality of life between inclusion and the end of self-hypnosis practice between the 2 groups of participant | week 16 after enrollment
  Quality of life will be evaluated by the SF-12 scale Score calculated with a software
Comparison between the 2 groups the care consumption between inclusion and the end of self-hypnosis practice | week 16 after enrollment
  The care consumption will collected on a patient diary.
Observance of self-hypnosis sessions at home | week 8 after enrollment
  Duration and localization of the session will be collected on a patient diary.
Observance of self-hypnosis sessions at home | week 16 after enrollment
  Duration and localization of the session will be collected on a patient diary.
Observance of self-hypnosis sessions at home | week 32 after enrollment
  Duration of the session will be collected on a patient diary.
Observance of self-hypnosis sessions at home | week 32 after enrollment
  Localization of the session will be collected on a patient diary.
Comparison of the variation of perceived stress between inclusion and the end of self-hypnosis practice between the 2 groups of participant | week 16 after enrollment
  Stress will be evaluated by the Perceived Stress Scale (PSS) min score = 10 and max score = 50 score < 27 : stress management by the person

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Reynaud, Principal Investigator — CHU de La Réunion
Locations (1):
- CHU de La Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reynaud D, Bruneau L. Feasibility and acceptance of self-hypnosis to reduce chronic stress levels on family in-home caregivers of elderly people: protocol for the POSSAID pilot, randomised, wait-list controlled trial. BMJ Open. 2022 Dec 30;12(12):e066749. doi: 10.1136/bmjopen-2022-066749. PMID 36585135